CLINICAL TRIAL: NCT01025557
Title: The Effects of Isovolumetric and Isocaloric Preloads of Various Types of Milk on Food Intake, Subjective Appetite and Glycemic Response in Healthy Young Men and Women
Brief Title: Isovolumetric and Isocaloric Preloads of Various Types of Milk on Food Intake, Subjective Appetite and Glycemic Response
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Dairy Farmers of Ontario (Other); Mondelēz International, Inc. (Industry); Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Milk Study - Experiment 1; DFO_24235
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Diabetes Prevention; Obesity Prevention
Keywords: Food intake; Blood glucose; Milk
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Chocolate milk (Experimental)
  Interventions: Other: Dietary intervention
- Milk (Experimental)
  Interventions: Other: Dietary intervention
- Infant formula (Experimental)
  Interventions: Other: Dietary intervention
- Soy beverage (Experimental)
  Interventions: Other: Dietary intervention
- Water (Experimental)
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — Dietary treatments with beverages

SUMMARY:
The purpose of this protocol is to study the effects of fluid milk products on satiety, food intake, and glucose metabolism in healthy young men and women. Experiment 1: The specific objective is to investigate isovolumetric amounts of milk (2% M.F.), chocolate milk (1% M.F.), a soy beverage, cow's milk-based infant formula, and water (control) on satiety and food intake and on blood glucose before and after a meal. A fixed volume approach is based on the commercially available serving size. Experiment 2 will examine equicaloric amounts of milk (2% M.F.), chocolate milk (1% M.F.), a soy beverage, cow's milk-based infant formula, a glucose drink and water (control) the treatments in order to investigate macronutrient composition on satiety and food intake and on blood glucose before and after the meal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non-smoking
* Aged 20-30 years
* Body mass index between 20 and 24.9 kg/m2

Exclusion Criteria:

* Diabetes
* Medication
* Lactose-intolerance or allergies to milk
* Breakfast skippers and those on an energy restricted diet

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Food intake | 30 minute

SECONDARY OUTCOMES:
Blood glucose | 0, 10, 20, 30, 50, 80, 110, 140 and 170 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Anderson, Ph.D., Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada